CLINICAL TRIAL: NCT03269812
Title: Laparoscopic Assisted Pull-through Versus Other Surgical Procedures for Treatment of Hirschsprung Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Hamada Takrouney, Principal investigator and Assistant lecturer of pediatric surgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: laparoscopy in Hirschsprung
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic operated group (Experimental): Under general anesthesia and insertion of ports for laparoscopic instruments, laparoscopic assisted mobilization of sigmoid colon and dissection till pelvis and removal of a ganglionic segment of colon and laparoscopic assisted pull through of colon then colo-anal anastomosis will be done,
  Interventions: Procedure: laparoscopic assisted pull-through oeration
- non laparoscopic operated group (Experimental): Under general anesthesia ,abdominal exploration ,removal of a ganglionic part by soav ,duhamel procedures and trans-anal pull through procedures.
  Interventions: Procedure: laparoscopic assisted pull-through oeration

INTERVENTIONS:
Procedure: laparoscopic assisted pull-through oeration — Under general anesthesia and insertion of ports for laparoscopic instruments, laparoscopic assisted mobilization of sigmoid colon and dissection till pelvis and removal of a ganglionic segment of colon and laparoscopic assisted pull through of colon then colo-anal anastomosis will be done,

SUMMARY:
To evaluate the outcomes of laparoscopic pull-through concerning constipation, incontinence and enterocolitis in comparison of other surgical procedures for treatment of Hirschsprung disease.

DETAILED DESCRIPTION:
Hirschsprung,s disease (HD) is a relatively common cause of intestinal obstruction in the newborn[1,2], The main goal in the treatment of patients with Hirschsprung,s disease is to resect the aganglionic segment and pull down the Normo-ganglionic bowel[3]. With the introduction of minimally invasive surgery, classic pull-through techniques were modified and improved with laparoscopy, because of the obvious advantages of laparoscopic-assisted pull-through operations in form of reduced pain and improved cosmoses this approach has gained much popularity[4,5].

ELIGIBILITY:
Inclusion Criteria:

1. Age from 6months to 3 years.
2. Both sexes.
3. Classic and long segment Hirshsprung.
4. Total a ganglionic colon.
5. Hirshsprung disease with leveling colostomy

Exclusion Criteria:

1. Patients <6 months and >3 years.
2. Short and Ultra-short Hirshsprung.
3. Recurrent cases of Hirshsprung.
4. Other contraindication of laparoscopy

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Constipation | from one to three months after operation
  persistace of inablilty to pass stool even after operation and treatment,it is physiological parameter and assisted by asking the mothers of patients about the bowel habits.

REFERENCES:
- [Background] Tomuschat C, Zimmer J, Puri P. Laparoscopic-assisted pull-through operation for Hirschsprung's disease: a systematic review and meta-analysis. Pediatr Surg Int. 2016 Aug;32(8):751-7. doi: 10.1007/s00383-016-3910-5. Epub 2016 Jul 1. PMID 27369964
- [Background] Taguchi T, Obata S, Ieiri S. Current status of Hirschsprung's disease: based on a nationwide survey of Japan. Pediatr Surg Int. 2017 Apr;33(4):497-504. doi: 10.1007/s00383-016-4054-3. Epub 2017 Jan 5. PMID 28058486